CLINICAL TRIAL: NCT01882036
Title: The Effects of Roux-en-Y Gastric Bypass on Mitochondrial Dysfunction and Type 2 Diabetes Mellitus
Brief Title: Bariatric Surgery And Adipose Inflammation Dysfunction and Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SURG-2018-26725
Record Dates: First submitted 2012-06-21; First posted 2013-06-20 (Estimated); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Type 2 Diabetes Mellitus; Insulin Resistance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gastric Bypass w/ matched hypocaloric diet (Active Comparator)
  Interventions: Procedure: Gastric Bypass w/ matched hypocaloric diet
- Hypocaloric Diet (Active Comparator)
  Interventions: Other: Hypocaloric diet

INTERVENTIONS:
Procedure: Gastric Bypass w/ matched hypocaloric diet — Roux en Y Gastric Bypass with Hypocaloric liquid diet for 10 days
  Arms: Gastric Bypass w/ matched hypocaloric diet
Other: Hypocaloric diet — Hypocaloric liquid diet for 10 days
  Arms: Hypocaloric Diet

SUMMARY:
The focus of this proposal is to define the mechanism by which bariatric surgery acutely improves insulin sensitivity. Our central hypothesis is that drastically reduced caloric intake early after Bariatric surgery improves the pro-inflammatory profile of macrophages, which in turn improves insulin sensitivity and glucose homeostasis.

DETAILED DESCRIPTION:
Bariatric surgery quickly improves tissue specific insulin sensitivity. Changes in glucose metabolism are seen within days after surgery, prior to any significant weight loss--raising the question of a difference between dietary restriction and early food intake after surgery. A major factor in the development of insulin resistance is obesity. It has been noted that by 3 months following Roux-en Y gastric bypass surgery in obese patients with (T2DM), fasting glucose and insulin levels are improved independent of weight loss, insulin resistance in muscle is lowered, and that the pro-inflammatory profile of resident microphages is lowered improving insulin sensitivity.

The focus of this proposal is to define the mechanism by which bariatric surgery improves impacts insulin sensitivity. Our long-term goal is to correlate these changes with direct measures of adipose tissue insulin resistance to develop novel immunotherapies towards reducing insulin resistance without surgery.

Our central hypothesis is that gastrointestinal rearrangement by various mechanisms impacts adipose tissue and improves the pro-inflammatory profile of macrophages improving insulin sensitivity and glucose homeostasis. To test this hypothesis we propose the following aims:

Specific Aim 1. Recruit a patient population and measure insulin sensitivity using homeostatic model assessment (HOMA) to measure insulin resistance (IR), cytokines, incretins, and serum adipokines in morbidly obese patients • prior to and 7-10 days following bariatric surgery while on a hypocaloric diet (surgery group) and •prior to and 7-10 days while following hypocaloric diet similar to bariatric surgery (diet group). Subjects will be assigned to the two arms; subjects assigned to the hypocaloric diet may be offered bariatric surgery after completion of the diet.

Specific Aim 2.

* Profile inflammatory macrophages, T cells and secreted factors in subcutaneous and visceral adipose tissue of patients prior to and following RYGB and hypocaloric diet treatments. • prior to and 7-10 days following surgery
* prior to and 7-10 days following hypocaloric diet similar to bariatric surgery

Specific Aim 3.

Assess the effects of bariatric surgery on ROS (reactive oxygen species) production, expression of transcription factors and enzymes of mitochondrial biogenesis, tissue FABP4, and biomarkers of oxidative stress and protein carbonylation in patients prior to and following surgery and in control diet subjects maintained on hypocaloric diet.

Specific Aim 4.

Determine the impact of bariatric surgery on lipolysis and the role of TLQP-21 (a genetically derived peptide that increases energy expenditure and prevents the early phase of diet-induced obesity).

ELIGIBILITY:
Inclusion Criteria::

1. Candidate for RYGB gastric bypass with insurance approval.
2. Willing to accept randomization to either immediate surgery, or delayed surgery after diet study.
3. Willing to undergo two sessions of testing before, and ten days after surgery (or initiation of dietary intervention).
4. BMI 35-45kg/m2
5. Pre-diabetes (ADA criteria) or T2DM with HbA1c< 8%.

Exclusion criteria:

1. T1DM.
2. Serious illness such as cancer, active chronic infection, cardiovascular disease greater that New York Heart Association class 2, chronic renal failure, chronic lung disease.
3. Inflammatory or celiac intestinal disease.
4. Untreated thyroid disease.
5. Serious psychiatric disease.
6. Excessive alcohol use.
7. Illicit drug use. -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2018-07-10 (Actual); Study Completion 2018-07-10 (Actual)

PRIMARY OUTCOMES:
Measure homeostasis model assessment i.e. estimated change in insulin resistance (HOMA-IR) index | Seven days before and 10 days following RYGB or hypocaloric diet similar to RYGB patients

CONTACTS AND LOCATIONS:
Overall Officials: Sayeed Ikramuddin, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States